CLINICAL TRIAL: NCT02887339
Title: Ethical, Legal, and Social Issues Substudy in Relation to the Genotype-Tissue Expression Project
Brief Title: Ethical, Legal, and Social Issues Substudy in Relation to the GTEx Project
Acronym: ELSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Laura Siminoff, Dean, College of Health Professions and Social Work, Temple University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10XS170
Record Dates: First submitted 2015-12-17; First posted 2016-09-02 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Standard Training; Online Training
Keywords: Informed Consent; Research donation request; Effective Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Tissue requesters from participating OPOs are randomly assigned to complete additional informed consent training through an interactive online training website.
  Interventions: Other: Training Website
- Control Group (Experimental): The control group of tissue requesters receive the standard training offered by their OPO and GTEx partners.
  Interventions: Other: Control

INTERVENTIONS:
Other: Training Website — Additional training website can be found at gtextraing.org
  Arms: Intervention Group
Other: Control — Standard training given by OPOs and GTEx staff
  Arms: Control Group

SUMMARY:
The Ethical, Legal and Social Issues Substudy in relation to the Genotype Tissue Expression Project (GTEx) aims to describe tissue requesters' approach to discussions about donation to GTEx and to assess the determinants of families' and patients' willingness to donate to GTEx. It also explores ethical issues such as privacy, risks, and release of incidental findings and recommend best practices for conducting authorizations and training requesters.

DETAILED DESCRIPTION:
The Genotype Tissue Expression Project (GTEx) is a partnership between multiple NIH agencies and funded by the Common Fund. Families who agreed to donation of organs and tissues for transplantation were asked to authorize the collection of additional tissues for GTEx by participating Organ Procurement Organizations (OPO). Donated tissues are placed in a National Cancer Institute biobank, and the donor's genome and medical record information analyzed and released to researchers through NIH's database of Genotypes and Phenotypes (dbGaP). The tissues and information will be kept in the biobank indefinitely and cell lines may be developed from the donated skin and blood.

An ethical, legal and social issues (ELSI) sub-study examines the issues surrounding risks to privacy and breach of confidentiality to family decision makers (FDM) as well as FDM perspectives on the return of findings to donor families. The ELSI sub-study assessed the authorization process and make suggestions for its improvement. Semi-structured interviews were completed with families who decided to donate to GTEx as well as those who refused to donate to the project. Tissue requesters (TR) who make the GTEx approaches for participating OPOs, were also asked to complete an online survey for each approach they completed for GTEx.

The study builds on this research team's extensive work in organ and tissue donation and the work currently being conducting during the ELSI pilot of the GTEx project. Specifically, the investigators propose to examine the impact of stress and complex information on donor families' decision-making to inform the consent process; understand how variations in requesters, consent approaches, and the characteristics of family decision makers affect understanding, recall of and willingness to donate tissues for research; consider the ethical and legal issues of the request and consent process; and, test a novel intervention designed to train tissue requesters to employ effective communication techniques when making requests for tissue. The overall goal is to develop a set of recommendations that will maximize the likelihood that family decision makers (FDM) make informed donation decisions under stressful circumstances. The specific aims of the ELSI GTEx study are:

This study will build on this research team's extensive work in organ and tissue donation and the work they are currently conducting during the ELSI pilot of the GTEx project. Specifically, the investigators propose to examine the impact of stress and complex information on the decision making of donor families to inform the consent process, understand how variations in requesters, consent approaches, and the characteristics of family decision makers affect understanding and recall of and willingness to donate tissues for research, consider the ethical and legal issues of the request and consent process, and test an intervention to train tissue requesters to employ effective communication techniques when making requests for tissue. The overall goal is to develop a set of recommendations that will maximize the likelihood that family decision makers (FDM) make informed donation decisions under stressful circumstances. The specific aims of the ELSI GTEx study are:

1. Identify elements of nonverbal and relational communication impacting FDM knowledge, recall and GTEx decision making. Using the methods and procedures of the pilot study, the investigators will conduct an observational study of the GTEx request process to understand the communication-related variables impacting FDM knowledge, recall and decision making. In addition, a subsample of audiotapes will be obtained from tissue-only donors whose consent conversations are conducted by telephone and are audiotaped. This will provide information about the important nonverbal and relational elements of communication on the outcome variables.

   H1a. Sociodemographic characteristics of FDM will impact the major outcomes of interest to this study (recall, comprehension and consent). Specifically, FDM who have more education, are white, female and younger will be more likely to donate, have better recall and knowledge.

   H1b. Relational elements of communication, such as confirmational messages (e.g., messages that expressed validation or acceptance) or persuasive tactics such as credibility, altruism, or esteem, and engaging in a lengthier conversation will be associated with a greater likelihood to donate have better recall and knowledge.

   H1c. Tissue requesters' and FDMs' comfort speaking about GTEx, the proclivity of FDMs to ask question and engage more proactively in the conversation will be associated with a greater likelihood to donate have better recall and knowledge.
2. Conduct a study, using a quasi-experimental design, to understand the impact of the stressful environment in which the requests occur. This study will assist the ELSI team to obtain an evidence base that will allow us to disentangle the effects of stress from the complexity of the information about the purpose of the donation and guide recommendations for a final consent process.
3. Adapt and test a communication intervention targeting tissue requesters' (TR) use of effective, ethically acceptable techniques that maximize the likelihood of consent.

H3a. Post intervention, TRs will exhibit more relational communication with FDMs during requests. H3b. Post intervention, TRs will spend more time attending to the emotional needs of FDMs.

H3c. Post intervention, TRs will spend more time discussing information identified as important to informed decision making for tissue donation.

H3d. Post intervention, there will be overall higher consent rates for donation to the research.

ELIGIBILITY:
Inclusion Criteria:

Participants must either be a:

1. family decision maker approached to donate their loved one's tissues to the GTEx project or
2. a staff person at an OPO that approaches family decision makers for the GTEx project.

Exclusion Criteria:

1. Persons who neither approached for GTEx or were approached are excluded from participation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2013-03; Primary Completion 2016-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of family members who chose to donate to GTEx | Up to 8 months after donation request
  Number of family decision makers who choose to donate to GTEx

SECONDARY OUTCOMES:
Knowledge and Comprehension of Elements of Consent | Up to 8 months after donation request
  Knowledge and comprehension were assessed by participant answers to questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Siminoff, PhD, Principal Investigator — Temple University; Heather Traino, PhD, Principal Investigator — Temple University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GTEx Consortium. The Genotype-Tissue Expression (GTEx) project. Nat Genet. 2013 Jun;45(6):580-5. doi: 10.1038/ng.2653. PMID 23715323